CLINICAL TRIAL: NCT06523088
Title: A Phase 1a Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Immunogenicity of PN20 in Healthy Adult Volunteers
Brief Title: A Study of PN20 in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chongqing Peg-Bio Biopharm Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2021-PK-PN20-32
Record Dates: First submitted 2024-07-22; First posted 2024-07-26 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2024-07

CONDITIONS: Chemotherapy-induced Thrombocytopenia; Immune Thrombocytopenic Purpura
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: It is an open-label study at first dose level, and switched to double-blind study starting from the second dose level.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PN20 group (Experimental): subcutaneous injections, a single dose
  Interventions: Drug: PN20
- Placebo group (Placebo Comparator): subcutaneous injections, a single dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PN20 — Six dose levels of PN20 will be evaluated
  Other Names: thrombopoietin receptor agonist
  Arms: PN20 group
Drug: Placebo — Placebo of PN20
  Arms: Placebo group

SUMMARY:
The main aim of this clinical trial is to assess the safety of PN20 in healthy volunteers aged 18 to 50 years. The main questions it aims to answer are:

* Is PN20 safe in adult? Researchers will compare PN20 to a placebo (a look-alike substance that contains no drug) to see if PN20 is safe.

Participants will

* Receive a single dose injection of PN20 or placebo according to weight,
* Stay in hospital for assessment.

DETAILED DESCRIPTION:
This is a single center, randomized, double-blind, placebo-controlled, dose escalation phase 1 clinical study, aiming to evaluate the efficacy, safety, immunogenicity and pharmacokinetic of PN20 in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female subjects aged 18 to 50 years;
2. Body mass index between 19.0-28.0 (inclusive), body mass index (BMI) = weight (kg)/height^2 (m^2);
3. Female subjects of childbearing age with negative serum pregnancy test results;
4. Platelet counts during the screening period and one day before enrollment are within the range of 100-300×10^9/L;
5. Eligible subjects of fertility must agree to use effective contraceptive measures or abstain from sex within 6 months after receiving the investigational drug;
6. Be able to understand and comply with the requirements of the protocol and expected to complete the entire trial process;
7. Voluntarily participate and sign the informed consent form.

Exclusion Criteria:

1. Abnormal results of vital signs examination with clinical significance determined by the investigator;
2. Positive test results for HIV-Ab, HCV-Ab, HBsAg, HBeAg, or treponema pallidum antibodies;
3. Abnormal results of laboratory test (blood routine, urine routine, blood biochemistry, coagulation) with clinical significance determined by the investigator;
4. Abnormal electrocardiogram with clinical significance or prolonged QT/QTc interval is, such as QTcB ≥ 430ms (male), or QTcB ≥ 450ms (female) (machine reading results); family history of QT prolongation;
5. Positive drug abuse test or alcohol test ≥20mg/dL;
6. Abnormal results of chest CT or COVID-19 screening (nucleic acid and C-reactive protein) with clinical significance determined by the investigator;
7. Have taken any drugs (including prescription drugs, over-the-counter drugs and Chinese herbal medicines) within 4 weeks before enrollment, except for external drugs that are not absorbed by the body;
8. Have used drugs known to cause significant damage to certain organs within 12 weeks before enrollment;
9. Participated, enrolled and been administered in other clinical trials within 3 months before enrollment, or used this investigational drug or similar drugs;
10. Received live attenuated vaccines within 28 days before administration of the trial drug and/or received inactivated vaccines within 7 days before administration, and/or plan to receive vaccines during the trial;
11. Allergic constitution, or history of drug allergy, or history of allergy to the ingredients of this investigational drug;
12. Have a history of major surgery or a history of blood donation ≥200 mL within 12 weeks before enrollment or who plan to donate blood during the study;
13. Have a history of any serious clinical disease, including but not limited to diseases of the digestive system, cardiovascular system, respiratory system, urinary system, musculoskeletal system, endocrine system, neuropsychiatric system (such as epilepsy, dementia, etc.), blood system, and immune system And those with a history of metabolic abnormalities, deep vein thrombosis, thrombocytopenia, thrombocythemia, platelet dysfunction, etc.;
14. Smoke more than 5 cigarettes a day or have a history of alcohol abuse in the 6 months before enrollment, that is, drink more than 14 units of alcohol per week (1 unit = 12 ounces or 360mL of beer, 1.5 ounces or 45mL of hard liquor with 40% alcohol content, 5 ounces or 150mL of wine);
15. Drink more than 1L of strong tea, coffee and/or caffeinated beverages every day;
16. Cannot tolerate venipuncture blood collection or have a history of needle or blood fainting;
17. Lactating, pregnant or planning to become pregnant or conceive in the near future;
18. The investigator believes the subject would be unsuitable for participation in this clinical study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2022-06-16 (Actual); Primary Completion 2023-01-05 (Actual); Study Completion 2023-01-05 (Actual)

PRIMARY OUTCOMES:
Treatment-related Adverse Events | up to 15 days
  Number of participants with treatment-related adverse events during the study will be collected and the percentage of AE of different grades as assessed by CTCAE v5.0 will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Liyan Miao, Principal Investigator — The First Affiliated Hospital of Soochow University
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangshu, China